CLINICAL TRIAL: NCT07172620
Title: Safety and Effectiveness of No-touch Technique for Ascending Aorta in Minimally Invasive Cardiac Surgery Coronary Artery Bypass Grafting(MICS-CABG)
Brief Title: Safety and Effectiveness of No-touch Technique for Ascending Aorta in MICS-CABG
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Arota notouch of MICS-CABG
Record Dates: First submitted 2025-04-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Bypass Grafting; Off-pump Coronary Artery Bypass; Minimally Invasive Cardiac Surgery; Coronary Arterial Disease (CAD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exposure group (MICS-Notouch group): Patients enrolled underwent non-extracorporeal coronary artery bypass grafting under direct vision through a small left thoracotomy, including the use of LIMA (left internal mammary artery) + SVG (saphenous vein graft) multibranch bypass grafts.
  Interventions: Procedure: Non-extracorporeal multiple coronary artery bypass graft (CABG) performed under direct visualization through a small incision in the left side of the chest.
- Control group (OPCAB group): Patients enrolled underwent conventional median open-heart surgery with multiple coronary artery bypass grafting under off-pump circulation.
  Interventions: Procedure: Multi-branch coronary artery bypass grafting with conventional median open heart and off-pump circulation

INTERVENTIONS:
Procedure: Non-extracorporeal multiple coronary artery bypass graft (CABG) performed under direct visualization through a small incision in the left side of the chest. — Exposure group (MICS-Notouch group): Direct visualization non-extracorporeal coronary artery bypass grafting with a small left chest incision, including the use of LIMA (left internal mammary artery) + SVG (saphenous vein) multibranch bypass grafting.
  Groups: Exposure group (MICS-Notouch group)
Procedure: Multi-branch coronary artery bypass grafting with conventional median open heart and off-pump circulation — Control Group (OPCAB Group): Conventional median open multiple coronary artery bypass grafting with extracorporeal circulation.
  Groups: Control group (OPCAB group)

SUMMARY:
The goal of this single-center prospective cohort study is to compare perioperative safety metrics and follow-up survival analyses in patients receiving Minimally Invasive Cardiac Surgery Coronary Artery Bypass Grafting(MICS-CABG) and Off-Pump Coronary Artery Bypass(OPCAB). The main question it aims to answer is:

Is the bridge vessel patency rate of patients in the MICS-Notouch group noninferior to that of a saphenous vein bridge with conventional open-chest bypass?

Participants will be divided into two groups:

Exposure group (MICS-Notouch group): non-extracorporeal circulation multiple coronary artery bypass grafting surgery performed under direct visualization of a small incision in the left chest, including the application of LIMA (left internal mammary artery) + SVG (saphenous vein) multiple bypass grafting.

Control group (OPCAB group): conventional median chest opening, non-extracorporeal circulation multi-branch coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
STATUS OF THE STUDY: Coronary Artery Bypass Grafting (CABG) surgery and Percutaneous Coronary Intervention (PCI) are important methods to address myocardial ischemia in coronary artery disease. CABG surgery, with its internal mammary artery bridging, can achieve a patency rate of more than 90% at 5 years after the procedure, which is currently the gold standard for the treatment of coronary artery disease. Although with the development of drug-eluting stents, coronary spinning mill technology and FFR technology, the incidence of mid- and long-term major adverse cardiovascular and cerebrovascular events (MACCE) of PCI treatment has been greatly reduced, CABG surgery is still the first choice for patients with complex coronary artery disease, left main stem disease and diabetes mellitus and other high-risk patients. However, traditional CABG surgery requires splitting the sternum, which is highly traumatic compared with PCI treatment, and carries a high surgical risk for patients with advanced age and comorbidities, as well as the risk of non-healing of the sternum. Minimal Invasive Cardiac Surgery-Coronary Artery Bypass Grafting surgery (MICS-CABG surgery) can reduce surgical trauma, surgical blood transfusion, and shorten postoperative hospitalization due to the avoidance of sternum injury.

Due to space constraints, MICS-CABG surgery cannot apply a proximal anastomosis to the ascending aorta and requires the use of a special sidewall clamp to clamp the ascending aorta, which poses two potential risks: 1. In patients with calcification and thickening of the ascending aorta, clamping of the ascending aorta may cause rupture of the intimal plaque and dislodgement, which can lead to the risk of cerebral infarction and peripheral arterial embolism; 2. minimal incision In bypass surgery, the proximal anastomosis of the ascending aorta has a very low tolerance rate. Due to the deep location of the ascending aorta, the surgical field and operating space are limited, and the suture is extremely difficult, if the anastomosis process occurs in the case of vascular tear, anastomotic leakage, or dislodgement of the sidewall clamp, it will cause serious uncontrollable aortic bleeding, which may endanger the patient's life in a short period of time.

SIGNIFICANCE: The optimization of the MICS-CABG surgical protocol through this topic reduces the surgical risk and removes the obstacles for the promotion of this technology.

In order to solve the problem of proximal anastomosis of MICS-CABG surgery in patients with calcification of the ascending aorta and to reduce the difficulty and risk of surgery. In 2020, our center began to explore the minimally invasive bypass surgery of ascending aorta non-touch (No-touch) technology, which refers to the bypass surgery without any manipulation of the ascending aorta, the proximal anastomosis of the bridge vessel in the axillary artery, through the first intercostal space of the bridge vessel to the thoracic cavity for the distal continuation of the anastomosis. The advantages of this technique are: 1) avoiding ascending aortic manipulation eliminates the risk of cerebral infarction and peripheral arterial embolism caused by plaque dislodgement from the ascending aorta; 2) the axillary artery rarely exists in calcification, and the vascular condition is good; 3) the axillary artery is simple to reveal, with plenty of room for maneuvering, and it can be anastomosed under direct vision, which greatly reduces the difficulty of the procedure, and if the anastomosis bleeds after the completion of the anastomosis, the bleeding is simple to stop, which decreases the risk of surgical manipulation.

This study will evaluate the safety and efficacy of this technique in a prospective cohort study. If the safety and efficacy of this technique are confirmed to be good, it will greatly expand the indications of this cutting-edge technique of MICS-CABG, optimize the surgical plan, reduce the surgical difficulty and shorten the learning curve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angina pectoris who experience functional limitations in daily life and work despite conservative medical treatment and who require coronary artery bypass grafting surgery, as confirmed by coronary angiography, are eligible for enrollment.
* Patients with calcification of the ascending aorta, as confirmed by CT, who are not suitable for sidewall clamping are also eligible for enrollment.

Exclusion Criteria:

* The patient presents with an old, large myocardial infarction with no surviving myocardium, as evidenced by both isotope and echocardiographic imaging. This is a group of patients who are prone to complications, including significant cardiac enlargement, a cardiothoracic ratio greater than 0.75, an ejection fraction (EF) less than 30%, a left ventricular diameter (LVDd) greater than 70mm, the presence of a left ventricular ventricular wall tumor, or severe arrhythmia. Intraoperative hemodynamic instability;
* Valve surgery or other intracardiac surgery at the same time;
* Patients expected to undergo extracorporeal circulation surgery;
* Poor myocardial infarction conditions, extensive lesions, distal or full diffuse stenosis, or lumen diameter less than or severe calcification that cannot be anastomosed.
* Previous open heart surgery.
* Patients with preoperative hemodynamic instability requiring emergency surgery.
* Other conditions include terminal malignant tumors, uncontrollable infections, bleeding, persistent progressive degenerative systemic diseases, severe brain injuries, and multiple organ failure. Additionally, other significant organ function serious impairments, such as severe liver function impairment, severe heart failure, or cardiogenic shock, may also be considered contraindications. Inability to tolerate surgery may also be considered a contraindication.
* The participant declines to take part in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients to undergo coronary artery bypass grafting due to coronary heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Saphenous Vein Bridge Vessel Patency Rate | 1-14 days after surgery
  The patients' bridge vessel patency is assessed by angiography within 1-14 days after surgery.
Early Postoperative Saphenous Vein Bridge Vessel Patency Rate | 1-14 days after surgery
  The patients' bridge vessel patency is assessed by Coronary Computed Tomography Angiography within 1-14 days after surgery.

SECONDARY OUTCOMES:
Perioperative Safety Indicators | One year after surgery
  The following variables were considered: transfusion volume, extracorporeal circulation transfer rate, IABP and ECMO utilization rate, reoperation rate, incidence of poor wound healing, 1-year postoperative bridging vessel patency rate (CT or angiography), incidence of perioperative MACCE, incidence of atrial fibrillation, incidence of renal failure, incidence of re-tracheal intubation, duration of postoperative hospitalization, duration of ICU stay, duration of mechanical ventilation, and hospitalization costs.
Survival Analysis | One year after surgery
  The occurrence of MACCE (including all-cause mortality, re-bypass or stenting, acute infarction, and stroke), as well as readmission for infarction or heart failure at 1, 3, 6, and 12 months postoperatively, will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Yunpeng, PhD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided